CLINICAL TRIAL: NCT07066475
Title: A Registry-Based Cohort Study on the Clinical Outcomes of Spinal Cord Glioma Resection Via the Dorsolateral Sulcus Approach
Acronym: DLS
Status: Recruiting | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY2025-143-02
Record Dates: First submitted 2025-06-25; First posted 2025-07-15 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Spinal Cord Cancer; Spinal Cord Neoplasm; Spinal Cord Tumor
Keywords: Spinal Cord Glioma; Spinal Cord Astrocytes; Intramedullary tumor
MeSH Terms: conditions — Spinal Cord Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DLS Group: Patients who underwent tumor resection through the dorsolateral sulcus approach
- PMS Group: Patients who underwent tumor resection through the posterior median sulcus approach

SUMMARY:
Spinal cord gliomas are the most common type of primary intramedullary malignant tumors, with a low incidence and a peak onset age of approximately 35 years. They are slightly more prevalent in males than females. Clinical manifestations vary depending on tumor characteristics and location, typically presenting with axial pain and displaying a tendency for unilateral, infiltrative growth. Prognosis is generally poor, and effective treatment options are limited aside from surgical resection. Common surgical approaches for intramedullary tumor removal include the posterior median sulcus approach, the dorsolateral sulcus approach, and surface entry techniques.

Preliminary clinical observations suggest that the dorsolateral sulcus approach may offer superior preservation of neurological function and quality of life. However, due to limited research evaluating the safety and efficacy of different surgical routes, the traditional posterior median sulcus approach remains widely used.

This single-center, registry-based cohort study aims to compare the outcomes of spinal cord glioma resection via the dorsolateral sulcus approach versus the posterior median sulcus approach. Patients with laterally located tumors undergoing surgical treatment, classified according to the 2021 WHO criteria, will be included. Neurological function scores and quality-of-life assessments will be used to evaluate prognosis and survival, in order to determine the optimal surgical approach for spinal cord glioma resection.

DETAILED DESCRIPTION:
Spinal cord gliomas are rare primary intramedullary tumors characterized by lateralized infiltrative growth and limited treatment options beyond surgical resection. Due to the anatomical complexity and functional sensitivity of the spinal cord, the choice of surgical approach significantly impacts postoperative neurological outcomes.

The traditional posterior median sulcus (PMS) approach provides direct midline access for tumor removal but carries a considerable risk of damage to central neural tracts. The dorsolateral sulcus (DLS) approach offers an alternative route for laterally located tumors, potentially sparing critical midline structures and improving functional outcomes.

This single-center, registry-based cohort study aims to evaluate and compare the clinical outcomes of spinal cord glioma resections performed via the DLS and PMS approaches. Patients will be enrolled based on eligibility criteria including lateralized tumor growth confirmed by imaging and histopathology, in accordance with the 2021 WHO classification of CNS tumors.

Primary and secondary outcomes will be assessed using validated clinical scales, including:

Visual Analog Scale (VAS) for pain assessment McCormick Functional Grading Scale Japanese Orthopaedic Association (JOA) Score for spinal cord function SF-36 Health Survey for quality of life evaluation Functional assessment of posterior column integrity Outcome assessments will be performed at five scheduled time points: preoperatively, and postoperatively at 1 month, 3 months, 6 months, and at the last follow-up visit. The study will evaluate neurological recovery, extent of resection, tumor recurrence, postoperative complications, and overall survival. This research aims to identify the optimal surgical approach that maximizes tumor resection while preserving neurological function in patients with spinal cord gliomas.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 3 and 75 years
2. Undergoing surgical resection of spinal cord tumor
3. Histopathological diagnosis of spinal cord glioma based on routine pathological examination
4. Availability of complete clinical data and willingness to participate in follow-up
5. Informed consent obtained from the patient and/or legal guardians or immediate family members

Exclusion Criteria:

1. Age under 3 years or over 75 years
2. Receipt of radiotherapy, chemotherapy, or anti-tumor biological therapy within 1 month prior to enrollment
3. Receipt of immunotherapy within 3 months prior to enrollment
4. Participation in other clinical trials within 3 months prior to enrollment
5. History of severe allergic reactions or known allergy-prone constitution
6. Pregnant or breastfeeding women, or individuals of childbearing potential not using adequate contraception
7. Presence of other severe medical conditions or uncontrolled infections
8. History of drug abuse, substance misuse, chronic alcoholism, or HIV infection
9. Uncontrolled epileptic seizures or psychiatric disorders resulting in loss of self-control

Ages: 3 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is a single-center registry study including patients aged 3-75 years who were diagnosed with spinal cord glioma by histopathology and underwent surgical resection. All participants provided informed consent and were able to complete follow-up assessments.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Extent of resection | Preoperative MRI and MRI re-examinations conducted within 3 days after the surgery
  The extent of tumor resection was evaluated by comparing the preoperative and postoperative magnetic resonance images, and the criterion for judgment was that the tumor volume decreased by more than 50%.
Number of Participants with Preserved Dorsal Column Function (Assessed by clinical neurological examination and intraoperative electrophysiological monitoring ) | Preoperative, 1 month, 6 months
  Dorsal column function will be assessed through standardized clinical neurological examination, including evaluation of proprioception (joint position sense), vibration sense, and gait. Dysfunction is defined as the presence of generalized numbness or painful dysesthesias below the surgical level, accompanied by proprioceptive loss and/or gait disturbance. * This definition is based on previously published clinical criteria for dorsal column dysfunction in patients with intramedullary spinal cord tumors, as described by Manzano et al.
Pain Level (VAS Score) | Preoperative, 1 month postoperative, 6 months postoperative, and 12 months postoperative
  Assessment of pain severity using the Visual Analog Scale (VAS), with scores ranging from 0 (no pain) to 100 (worst possible pain).
Neurological Functional Status (McCormick Grade) | Preoperative, 1 month postoperative, 3 months postoperative, 6 months postoperative, and 12 months postoperative
  Evaluation of neurological status using the McCormick Functional Grading Scale to compare surgical approaches. The scale ranges from Grade I (normal gait and function) to Grade IV (severe disability or paraplegia).

SECONDARY OUTCOMES:
SF-36 quality of life metrics | 6 months and 12 months postoperative
  Quality of life will be assessed using the 36-Item Short Form Survey (SF-36), a validated questionnaire that evaluates multiple health domains including physical functioning, bodily pain, general health, vitality, social functioning, emotional role, and mental health. Each domain is scored from 0 to 100, with higher scores indicating better health-related quality of life.
Progression-Free Survival (PFS) | From date of surgery until tumor progression or death, assessed up to 24 months
  Progression-free survival is defined as the time from surgery to the first documented tumor progression or death from any cause. Progression is determined by imaging and/or neurological deterioration.
Overall Survival (OS) | From date of surgery to death from any cause, assessed up to 36 months
  Overall survival is defined as the time from surgery to death from any cause. Survival status will be monitored through clinic visits or follow-up contact.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Neurosurgical Institute, Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to share de-identified individual participant data including baseline characteristics, treatment assignment, primary and secondary outcome measures. Additionally, the investigators will provide the study protocol, data dictionary, and statistical analysis plan. Data will be shared in a secure format to protect participant confidentiality.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Start date: Within 6 months after study completion and publication of results. End date: 5 years after the start date.
Access Criteria: Access to the de-identified individual participant data (IPD) and supporting documents will be granted only to qualified researchers who submit a formal request describing their research purpose. Requests will be reviewed by the study team for approval. Approved applicants will be required to sign a data use agreement before receiving access. Data will be shared through a secure platform to ensure confidentiality and proper use.
URL: https://www.ncrcnd.org.cn/